CLINICAL TRIAL: NCT03354975
Title: Dissemination of Exposure-Based Treatment for Anxiety: Experiential Training for Community Therapists
Brief Title: Experiential Training for Community Therapists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 260359; F31MH112211 (NIH)
Record Dates: First submitted 2017-11-13; First posted 2017-11-28 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiential Training (Experimental)
  Interventions: Behavioral: Experiential Training
- Training-as-usual (Active Comparator)
  Interventions: Behavioral: Training-As-Usual

INTERVENTIONS:
Behavioral: Experiential Training — Participants in the experiential training will be provided with information about using exposure therapy to treat patients with anxiety via lecture-style teaching. Then, they will themselves undergo a one-session phobia treatment for spiders.
  Arms: Experiential Training
Behavioral: Training-As-Usual — The training-as-usual condition will incorporate passive and active learning components. The first half of the training will include lecture-style teaching about using exposure therapy to treat patients with anxiety. The second half of training will incorporate active learning components (e.g., role plays) to reinforce concepts discussed in the first half of training.
  Arms: Training-as-usual

SUMMARY:
The primary goal of this study is to evaluate the feasibility and acceptability of employing an experiential training approach that targets community mental health therapists' attitudes toward and use of exposure therapy. In addition to assessing attitudes and use of exposure therapy, the study will evaluate the feasibility of recruitment, randomization, retention, and assessment processes, as well as the acceptability of the experiential training relative to training-as-usual. To assess these outcomes, community therapists will be randomized to experiential training or training-as-usual. A subset of therapists from each arm will also complete qualitative interviews to further assess acceptability of the training approaches. The training-as-usual condition will include a traditional one-day workshop that focuses on principles of exposure and incorporates active learning strategies. The experiential training will include a one-day workshop that teaches principles of exposure and has therapists themselves undergo a one-session phobia treatment for spiders. Therapists in both training conditions will be asked to attend weekly consultation phone calls for a three-month period following the trainings.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be aged 21 and older with degrees (masters or doctorate) in a mental health field. They must be working in a community mental health clinic, currently treating at least one client with anxiety, and planning to continue providing therapy to at least one client with anxiety for the duration of the study. Participants must be interested in participating in a training workshop and able to commit to the time requirements for study completion. They must also be willing to provide an email or mailing address to complete study-related surveys. Finally, they must be able to read and speak English.

Exclusion Criteria:

* Participants cannot have previously attended a full day (8+ hours) workshop on exposure-based treatments for anxiety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Therapist Beliefs about Exposure Scale (TBES) at 3-month follow-up | Pre-training; 3-month follow-up
  The Therapist Beliefs about Exposure Scale is a 21-item self-report measure that assesses therapists' negative beliefs about exposure therapy. Agreement with each item is rated on a 5-point scale ranging from 0 (disagree strongly) to 4 (agree strongly), yielding a total score ranging from 0 to 84. Higher scores indicate more negative beliefs about exposure.
Change from baseline Exposure Therapy Clinical Use Survey (ETCUS) at 3-month follow-up | Pre-training; 3-month follow-up
  The ETCUS measures therapist-reported use of nine exposure therapy procedures, such as providing the rationale for exposure therapy, creating a hierarchy, and completing in-vivo exposures.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States